CLINICAL TRIAL: NCT04440319
Title: A 12-Week Double-Blind of Diabetes Nutrition Education in T2D
Brief Title: Diabetes Nutrition Education With Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andalas University (Other)
Collaborators: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, ICE YOLANDA PURI, Principle Investigator, Andalas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Andalas U
Record Dates: First submitted 2020-05-01; First posted 2020-06-19 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Type2 Diabetes Mellitus
Keywords: DNE mddule; Glycemic control; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study has a DM nutrition education module that will be determined to intervention group (individual with T2DM). While control group follow the conventional DM counseling.
Who Masked: Participant
Masking Description: Individual with T2DM in both of groups will not know their groups (single blind), but the researcher knows
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention groups (4 PHC/clinics) (Experimental): Intervention group are individual with T2DM who will receive DM nutrition counseling at selected Public Health Care (PHC). There are 75 subjects in Intervention group at selected 2 districts by randomly and 4 PHC which is selected based on cluster. DM nutrition counseling will be delivered by a selected nutritionist at each PHC. Nutritionist will educate the subjects following DM nutrition education module properly. DM nutrition education will be delivered for 3 months and 30 minutes for each meeting.
  Interventions: Behavioral: Intervention group
- Control groups (4 PHC/clinics) (Experimental): As the same with intervention group, the control group will have 75 subjects but at the different districts and PHC to avoid contaminant. Control group will follow conventional DM nutrition education. Therefore, there is a selected nutritionists will deliver DM counseling at each PHC.
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Intervention group — Intervention group is individual with T2DM who will receive DM Nutrition education for 3 months. There are 75 subjects in Intervention group at 2 districts and 4 Public Health Care (PHC).

SUMMARY:
T2DM in Indonesia has increased dramatically from 7.0% in 2017 to 10.9% in 2018. In Padang, West Sumatra, diabetes prevalence was 1.3% in 2013 and increased slowly in 2018. Majority of T2DM were not able to achieve optimal glycaemic glucose control measured using HbA1c with a target of less than < 6.5% based on WHO recommendation.

Problem Statement NCD guidelines provided management DM in general. Pedoman Gizi Seimbang was for healthy people. It is crucial to update the guideline following the current issues even the Indonesian consensus in 2015 provided a T2DM management diet.

Study Hypotheses There is a significant difference in glycemic control (HbA1c and FBG) nutritional status, knowledge, attitude, practice, quality of life, acceptability and adherence behavior among individuals with T2DM in intervention group.

Procedures Subjects will be divided into Intervention and control groups after they finished reading, signed a letter of agreement and informed consent. Subjects also have the right to be withdrawn after listening explanation of the investigators to seeking the potential participants based on inclusion criteria.

The individual with T2DM (intervention group) will follow the Diabetes Mellitus Nutrition Education (DNE) program based on the curriculum of DNE modules properly and certain measurements. There is a selected nutritionist at each PHC who will convey the DNE program. DM nutrition education counseling will be delivered every week for 30 minutes.

Individual with T2DM

* Baseline An individual with T2DM will be asked to fill the questionnaire and follow all of the measurements (Nutritional Status, Biochemical, Clinical, and Dietary Intake).
* Intervention (3 months) All of the subjects will follow the DM Nutrition Education program for 3 months which will be delivered by nutritionists in PHC.
* Follow up (3 months) All of the subjects will continue the program independently in 3 months. Then, the subjects will do the same activity as a baseline to compare the data between baselines, intervention and follow up Control The individual with T2DM in the control group will still follow the conventional DM nutrition education. After the DNE program finished, the material will also be distributed to the individual with T2DM in the control group.

DETAILED DESCRIPTION:
Phase I: Needs Assessment Research Design This is a descriptive statistics study and the aims are to determine the current practice of managing diabetes mellitus among nutritionists. The need for having DM nutrition education among individual with T2DM will be conducted following Cross-sectional study.

Subjects The need assessment will be conducted among all nutritionists at all PHC and individual with T2DM at selected PHC at Padang city.

Sampling The nutritionists will be recruited at all of PHC in Padang City and there are 50 nutritionists. PHC will be recruited using multiple random sampling among districts. Then, individual with T2DM will be selected using simple random sampling among selected PHC. One PHC will be selected at each district. Regarding sample size calculation use HbA1c Standard Deviation, the subjects can be gained, are 158. Therefore, 158 subjects are divided into 11 Districts. There are 12 T2DM patients that will be selected each selected PHC in every district using Random Block. Subjects will be selected following visiting individual with T2DM at PHC.

The study will be conducted at all Public Health Center (PHC) in Padang City. An individual with T2DM will be selected based on inclusion and exclusion criteria, multiply random sampling following a city (Padang), simple random sampling in every district and PHC. One PHC will be selected in every district following the highest number of T2DM patients in each district.

Statistical Analysis Descriptive statistics will be used to examine socio-demographic and current management among nutritionists. The need DM nutrition education among individual with T2DM data, the mean and Standard Deviation (SD) will be calculated for normally distributed continuous variables and frequency (f) and percentage (%) for nominal variables. Pearson's chi-square test will be used to examine independent variables.

Data Collection A Google form questionnaire will be developed and be done pre-test among nutritionists perspective. Pre-test questionnaires will be start at PHC outside Padang. Subjects will be taken 10 nutritionists at selected PHC. The items are Socio-demographic characteristics, Management of diabetes at PHC, Nutritional status measurement, DM education tools, current practice management T2DM, the need DM nutrition education, and DM of knowledge-attitude-practice level. The questionnaire will be distributed to all nutritionists using media social (what application). Data will be key in using the latest SPSS version.

A set questionnaire will be developed among individual with T2DM perspective to determine the need DM nutrition education at PHC. The questionnaire will be tested (pre-test) following selected subjects (10%) at a selected PHC in Padang. A selected PHC is different with 11 PHC that had been selected as simple random sampling accordingly.

Phase II: Development and Assessment Module

The module should be assessed following five expert panel review. Five expert panel reviews will assess the module using a set questionnaire.

The validity is to assess how well the idea of a theoretical construct is represented in a questionnaire. A good module should be analysed regarding the reliability and validity process that is a crucial part of a quantitative research inquiry. Therefore, the result can be studied on construct validity.

Face validity refers to researchers' subjective assessments of the presentation and relevance of the measuring instrument as to whether the items in the instrument appear to be relevant, reasonable, unambiguous and clear.

Content validity refers to whether the content of the questions or items measured in the instrument is representative and adequate when attempting to measure phenomena.

Construct validity is an important part of content validity which provides evidence of the degree of aspects and covariance. Hence, it can be representative of the targeted construct module.

The developing module will be continued with the assessment of the module. Actually, there were no decisions for the number maximum of expert panel review, however, at least five Experts panel will be evaluated and assessed the module. Expert panel reviews are Indonesian nutritionists, dietitians, researchers who are experts in nutrition.

To determine the content domain, the qualitative research method used a semi-structured in-depth interview with five expert panel reviews. The module should have content five items; module should reach population target, module content should be implemented precisely, the module should be delivered at the right time, the module should enhance behavior T2DM patients, and module content should alter T2DM patients self-concept in DM.

Following a validated questionnaire of Sidek Mohd and Jamaludin Ahmad in module content, the experts will determine the level of content DM nutrition education module. The range of scale for this assessment is from 1 (Extremely Agree) to 5 (Extremely Disagree).

A set DM nutrition education module curriculum module will be prepared to deliver the materials to the patients. The DM nutrition education will be developed based on Nutritionists and T2DM perspective on need assessment phase. DM nutrition education module was assessed among expert panel reviews. After that, the materials DM nutrition education module will be delivered by introducing DM, symptom, ethology, CHO counting and exchange, food recommendation, cooking method, reading food labeling, and exercise.

The curriculum will be conveyed in the class twice a month for 60 minutes. There will be materials that patients can bring at home and be practiced as a guideline.

The study is divided into intervention and control groups. After intervention finished, the material will also be distributed to T2DM patients in the control group. Furthermore, they will have the same knowledge after the Nutrition Education program finished. Actually, no differences module which will be delivered among groups. However, the timing to distribute the module should be considered to avoid the effect of a contaminant between groups.

The module will be prepared based on the result from a needs assessment in Phase I. Besides that, materials will follow Indonesian consensus, and guidelines, books that were released from the Indonesian Ministry of Health. The module should follow the management standard of the Indonesian Ministry of Health.

Phase III : Treatment and Evaluation Research Design This is a cluster Randomized Controlled Trial study. Implementation of module is to compare and determine effectiveness Nutrition Education Module diabetes mellitus between intervention and control groups. Data collection will be started from June 2020 to August 2020.

Sampling The clusters will be recruited by Puskesmas (PHC) and random by district will be selected following simple random sampling. Districts are selected based on the highest number of T2DM patients. Therefore, there are four clusters in each group and there are two districts each groups. The districts in intervention group are Kuranji and Pauh and the control group are Padang Selatan and Padang Utara. PHC (clusters) in the intervention group are Kuranji, Belimbing, Ambacang, and Pauh. PHC in the control group are Seberang Padang, Rawang Barat, Alai, and Air Tawar.

Sample Size Number of sample of each arm using 2 groups means comparison is n1 = 36, number of cluster, size (m) is m=4, number of sample size per cluster is n2 = 41 and Total sample is n2 = 75. Using α=0.05, power = 80%, ICC =0.05, total sample are 150 with 75 subject per arms.

Data will be collected using questionnaire with 5 sections. They are Section A: Socioeconomic and Demographic Data, Section B: Glycaemic control, Section C: Nutritional Status, Lipid Profile, and Blood Pressure, Section D: Knowledge, Attitude, Practice, and Section E: Quality of Life.

Individual with T2DM (intervention group) will follow Diabetes Mellitus Nutrition Education (DNE) program based on the curriculum of DNE modules properly and certain measurements. There is a selected nutritionists at each PHC who will convey the DNE program. DM nutrition education counselling will be delivered every week for 30 minutes. Before the DNE is started, selected nutritionists will be introduced of DNE program and curriculum to avoid misunderstanding during the program running.

In order to avoid contamination among groups, nutritionists (intervention group) will be asked to fill in the inform consent and be informed to not show the DM Nutrition Education Module and tool kits to subjects in the control group.

Individual with T2DM in control group will still follow the convention DM nutrition education. After DNE program finished, the material will also be distributed to individual with T2DM in the control group. Furthermore, they will have the same knowledge when the program finished. Actually, there is no differences module which will be distributed among groups. However, the timing to distribute the module should be considered to avoid the contaminant between groups

Data Analysis Statistical analyses will be performed using the latest version of STATA. The data will be checked for normality. Missing treatment intervention data for 3 months (three) and follow up 3 (three) months using an Intention-to-treat (ITT) will be implemented. Baseline data are missing when a mean imputation procedure is done.

Descriptive statistics will be expressed as portions, mean (SD). Time trend for treatment effect will be estimated from General Linear Model (GLM). GLM is to determine the between-group difference at 3 months intervention and 3 months follow up.

Differences between baseline, treatment 3 (three) months and 3 (three) months follow up will be calculated for each outcome. Estimation within and between intervention and control groups will be tested using two way-ANOVA. Sociodemographic characteristic data will be expressed as proportions, mean and Standard Deviation (SD).

One-way repeated measured ANOVA is to test independent variable and a continuous (interval or ratio) dependent variable (within groups). Then, two-way repeated measured ANOVA to test independent variable and dependent variable between groups. However, if the relationship between the covariate and the dependent variable is not linear, ANCOVA is inappropriate.

ELIGIBILITY:
Inclusion Criteria:

* T2DM Patients with new diagnosed at least 6 months
* Patients with range age 18-65 years old
* Male and female who can read and write
* Patients can communicate well

Exclusion Criteria:

* T2DM patients with stroke and complication
* T2DM patients who are pregnant and breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and Female
Enrollment: 150 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
HbA1c and Fasting blood glucose | 3 months
  HbA1c will be analyzed using high performance liquid chromatography, D-10. 158 subjects will be asked to fasting before fasting blood glucose measurement, which will be undertaken by trained clinical staff.
Statistical analyses for HbA1c and Fasting blood glucose | 3 months
  Statistical analyses will be performed using the latest version of STATA. The data will be checked for normality. Descriptive statistics will be expressed as portions, mean (SD). The time trend for the treatment effect will be estimated from the General Linear Model (GLM). GLM is to determine the between-group difference at 3 months intervention. Differences between baseline, treatment 3 (three) months will be calculated for each outcome. Estimation within and between intervention and control groups will be tested using two way-ANOVA. Sociodemographic characteristic data will be expressed as proportions, mean and Standard Deviation (SD). One-way repeated measured ANOVA is to test the independent variable and a continuous (interval or ratio) dependent variable (within groups). Then, two-way repeated measured ANOVA to test the independent variable and dependent variable between groups.

SECONDARY OUTCOMES:
Blood Pressure | 3 months
  Blood pressure (mm Hg) will be measured following Indonesian consensus 2015. They divides into Systolic < 140mmHg and Diastolic <90mmHg.
Statistical analyses for Blood Pressure | 3 months
  Statistical analyses will be performed using the latest version of STATA. The data will be checked for normality. Descriptive statistics will be expressed as portions, mean (SD). The time trend for the treatment effect will be estimated from the General Linear Model (GLM). GLM is to determine the between-group difference at 3 months intervention. Differences between baseline, treatment 3 (three) months will be calculated for each outcome. Estimation within and between intervention and control groups will be tested using two way-ANOVA. Sociodemographic characteristic data will be expressed as proportions, mean and Standard Deviation (SD). One-way repeated measured ANOVA is to test the independent variable and a continuous (interval or ratio) dependent variable (within groups). Then, two-way repeated measured ANOVA to test the independent variable and dependent variable between groups
Body Mass Index (BMI), assessed by Seca-Tanita scale | 3 months
  BMI (kg/m2) will be measured by Seca - Tanita scale. Indonesian consensus 2015 divides Body Mass Index (BMI) for T2DM become : BMI underweight (<18.5);BMI normal (from 18.5 to 22.9);BMI overweight (≥23.0);BMI with the risk of overweight (23.0- 24.9);Obesity I (25.0 - 29.9);Obesity II (≥30).
Statistical analyses for Body Mass Index (BMI) | 3 months
  Statistical analyses will be performed using the latest version of STATA. The data will be checked for normality. Descriptive statistics will be expressed as portions, mean (SD). The time trend for the treatment effect will be estimated from the General Linear Model (GLM). GLM is to determine the between-group difference at 3 months intervention. Differences between baseline, treatment 3 (three) months will be calculated for each outcome. Estimation within and between intervention and control groups will be tested using two way-ANOVA. Sociodemographic characteristic data will be expressed as proportions, mean and Standard Deviation (SD). One-way repeated measured ANOVA is to test the independent variable and a continuous (interval or ratio) dependent variable (within groups). Then, two-way repeated measured ANOVA to test the independent variable and dependent variable between groups.
Knowledge-Attitude-Practice DM questionnaire | 3 months
  Knowledge-Attitude-Practice DM questionnaires are adapted from Besher Gharaibeh, Fatema et al and Indonesian Ministry of Health questionnaire. There are 17 knowledge questionnaires, 25 attitude questionnaires, and 7 practices questionnaires.
  Knowledge The knowledge categorical will be divided into high, moderate, and low level. The high score is 14-17, the moderate score is 7-13, and the lowest score is 0-6.
  Attitude The highest score is 43-125, the moderate score is 26-42, and the lowest score is 0-25
  1 = Do not extremely agree 2= Do not agree 3 = Not sure 4 = Agree 5 = extremely agree Practice The practice categorical will be divided into high, moderate, and low level. The high score is 6-7, the moderate score is 3-5, and the lowest score is 0-6.
Statistical analyses for knowledge-attitude-practice DM | 3 months
  Statistical analyses will be performed using the latest version of STATA. The data will be checked for normality. Descriptive statistics will be expressed as portions, mean (SD). The time trend for the treatment effect will be estimated from the General Linear Model (GLM). GLM is to determine the between-group difference at 3 months intervention. Differences between baseline, treatment 3 (three) months will be calculated for each outcome. Estimation within and between intervention and control groups will be tested using two way-ANOVA. Sociodemographic characteristic data will be expressed as proportions, mean and Standard Deviation (SD). One-way repeated measured ANOVA is to test the independent variable and a continuous (interval or ratio) dependent variable (within groups). Then, two-way repeated measured ANOVA to test the independent variable and dependent variable between groups.
Quality of life, assessed by DM Quality of Life questionnaire | 3 months
  There are 16 quality of life DM question, is adapted from Singh as previous studies, and following Likert scale.
  The highest score is 28-80, the moderate score is 17-27, and the lowest score is 0- 16
  1 = not extremely satisfied 2= not agree satisfied 3 = Not sure 4 = satisfied 5 = extremely satisfied
Statistical analyses for quality of life | 3 months
  Statistical analyses will be performed using the latest version of STATA. The data will be checked for normality. Descriptive statistics will be expressed as portions, mean (SD). The time trend for the treatment effect will be estimated from the General Linear Model (GLM). GLM is to determine the between-group difference at 3 months intervention. Differences between baseline, treatment 3 (three) months will be calculated for each outcome. Estimation within and between intervention and control groups will be tested using two way-ANOVA. Sociodemographic characteristic data will be expressed as proportions, mean and Standard Deviation (SD). One-way repeated measured ANOVA is to test the independent variable and a continuous (interval or ratio) dependent variable (within groups). Then, two-way repeated measured ANOVA to test the independent variable and dependent variable between groups.
Waist Circumference (WC) | 3 months
  Waist Circumference (WC) is predictor parameter of T2DM. WC for man is ≥94 cm and for woman is Woman ≥ 80 cm.
Statistical analyses for Waist Circumference | 3 months
  Statistical analyses will be performed using the latest version of STATA. The data will be checked for normality. Descriptive statistics will be expressed as portions, mean (SD). The time trend for the treatment effect will be estimated from the General Linear Model (GLM). GLM is to determine the between-group difference at 3 months intervention. Differences between baseline, treatment 3 (three) months will be calculated for each outcome. Estimation within and between intervention and control groups will be tested using two way-ANOVA. Sociodemographic characteristic data will be expressed as proportions, mean and Standard Deviation (SD). One-way repeated measured ANOVA is to test the independent variable and a continuous (interval or ratio) dependent variable (within groups). Then, two-way repeated measured ANOVA to test the independent variable and dependent variable between groups.

CONTACTS AND LOCATIONS:
Overall Officials: ICE Y PURI, Principal Investigator — Andalas University
Locations (1):
- Ice Yolanda Puri, Padang, WEST Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
The planning are to do data collection in phase 1 among nutritionist and individuals with T2DM perspective. Then, it will be followed with developing module in phase 2, and intervention in phase 3.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Phase 1 is on June 2020 Phase 2 is on July and August 2020 Phase 3 is on September, October and November 2020
Access Criteria: Data will be conducted following questionnaire.

REFERENCES:
- [Result] Barakatun Nisak MY, Ruzita AT, Norimah AK, Kamaruddin NA. Medical nutrition therapy administered by a dietitian yields favourable diabetes outcomes in individual with type 2 diabetes mellitus. Med J Malaysia. 2013;68(1):18-23. PMID 23466761